CLINICAL TRIAL: NCT06885359
Title: A Post-market Study Evaluating Clinical and Safety Outcomes of Bipolar Hemiarthroplasty Using CoCrMo LOCK Bipolar Femoral Heads in Subjects with Hip Fracture
Brief Title: CoCrMo LOCK Bipolar Femoral Heads FU
Status: Not yet recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-46
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Femoral Fractures; Hip Arthropathy
Keywords: Femoral head; Partial Hip Arthroplasty
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CoCrMo LOCK bipolar femoral head implanted patient: Patients who underwent hip arthroplasty with CoCrMo LOCK bipolar femoral heads from 1at January 2023 onwards.

SUMMARY:
Study design: monocentric, retrospective, observational and post-market clinical study.

Purpose: To demonstrate the safety and performance of CoCrMo LOCK bipolar femoral heads. The eligible study population is represented by the entire population that underwent a hip replacement with CoCrMo LOCK bipolar femoral heads from 1st January 2023 onwards at the site in accordance with the indication for use of the product.

DETAILED DESCRIPTION:
The study is aiming to demoranstrate safety and performance of LOCK Bipolar femoral heads and will do it by considering the rate of revision of any prosthesis component and dislocation, by x-ray evaluation, by patient reported outcomes and walking/residential status. Patients are followed for 2 years after hemiarthroplasty and data are collected at 6 timepoints (pre-operative, intra-operative, at discharge, 4-months follow up, 12 months follow up and 24 months follow up).

ELIGIBILITY:
Inclusion Criteria:

* Displaced intracapsular hip fracture (Garden III-IV).
* Subjects underwent a Bipolar Hemiarthroplasty with a CoCrMo LOCK Bipolar femoral head as per their Indication For Use from January 1st, 2023, onwards.
* No concurrent joint disease at the time of the surgery.
* Absence of severe cognitive dysfunction demonstrated by 3 or more correct answers on the Pfeiffer test.
* Ability to ambulate independently with or without walking aids before surgery.
* Subject willingness to participate.

Exclusion Criteria:

* Undisplaced or minimally displaced intracapsular hip fracture (Garden I-II).
* Any CoCrMo LOCK Bipolar femoral head contraindication for use as reported in the current Instruction For Use.
* Pathological fracture secondary to malignant disease.
* Subjects with rheumatoid arthritis or symptomatic osteoarthritis.
* Previous treatment to the same hip for a fracture at the time of the surgery.
* Subjects who were deemed unsuitable for the surgical procedures by the anesthesiologist.
* Severe cognitive dysfunction or cognitive impairment demonstrated by 2 or less correct answers on the Pfeiffer test.
* Unable to walk before surgery (e.g., wheelchair or bed-ridden subjects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent partial hip arthroplasty with CoCrMo LOCK bipolar femoral heads from 1st January 2023 onwards
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the revision rate of CoCrMo LOCK Bipolar femoral heads at 24 months after surgery. | At 24 months after intraoperative visit

SECONDARY OUTCOMES:
Evaluation of the dislocation rate (including close reduction) in subjects with CoCrMo LOCK Bipolar femoral heads at 24 months after bipolar hemiarthroplasty | At 24 months after intraoperative visit
Evaluation of the revision incidence of any hip component for any reason at 24 months after bipolar hemiarthroplasty. | At 24 months after intraoperative visit
Evaluation of acetabular erosion (according to Baker classification) in subjects with CoCrMo LOCK Bipolar femoral heads at 12 months after Bipolar Hemiarthroplasty. | At 12 months after intraoperative visit
Assessment of Harris Hip Score (HHS) at 24 months after Bipolar Hemiarthroplasty with CoCrMo LOCK Bipolar femoral heads. | At 24 months after intraoperative visit
  The Harris Hip Score goes from 0 to 100, which is the best result.
Assessment of Oxford Hip Score (OHS) completed by subjects with CoCrMo LOCK Bipolar femoral heads at 24 months after Bipolar Hemiarthroplasty. | At 24 months after intraoperative visit
  The Oxford Hip Score goes from 0 to 48, with 48 being the best outcome
Assessment of Pain Likert-scale in subjects with CoCrMo LOCK Bipolar femoral heads at 24 months after Bipolar Hemiarthroplasty. | At 24 months after intraoperative visit
  The pain Likert-scale is a 6-point scale: - severe and spontaneous - severe when walking - tollerable - occurs after activity - light intermittent - no pain
Comparison between pre-operative and 4-month walking ability. | Performed at preoperative visit and 4months follow up visit
  Functional evaluation
  At the pre-operative time-point, the ability to walk is categorized in:
  * "able to walk without aids",
  * "able to walk using one walking aid",
  * "able to walk using two walking aids",
  * "able to walk using the walking frame"
  * "unable to walk" (wheelchair or bed-ridden subjects)
  At the 4-month post-operative time-point, the ability to walk is investigated is categorized in:
  * "maintained" (if the subject is able to walk independently as before, with aids if necessary)
  * "not maintained" (if the subject needs support from another person or uses a wheelchair or is bed-ridden)
Comparison between pre-operative and 4-month residential status. | Performed at preoperative visit and 4months follow up visit
  Daily habit
  At pre-operative timepoint, subjects are categorized as subjects that before the fracture were used to live:
  * at their own home (alone or with assistance),
  * in a sheltered home for independent people,
  * in a nursing home for people who need assistance with personal care.
  At 4-month post-operative timepoint, the residential status is categorised in:
  * maintained (if the subject is living in the same dwelling as before fracture),
  * not maintained (if the subject moved to a sheltered accommodation or a nursing home)

CONTACTS AND LOCATIONS:
Locations (1):
- Splošna bolnišnica Celje, Celje, Slovenia